CLINICAL TRIAL: NCT06530940
Title: Diagnostic Interest of the Buccal Schirmer Test in Xerostomia During Sjögren's Syndrome: XERODIAG
Acronym: XERODIAG
Status: Not yet recruiting | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Fatma Said, Associate professor, University Tunis El Manar
Other Study IDs: XERODIAG
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Sjogren's Syndrome; Xerostomia; Diagnosis
Keywords: xerostomia; sjogren's syndrom; salivary flow; oral schirmer test
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: consisting of 90 patients with SS and confirmed xerostomia by SF measurement (<0.1 ml/minute).
  Interventions: Diagnostic Test: Buccal Schirmer Test
- Group 2: consisting of 90 patients with SS and normal SF (≥0.1 ml/minute).
  Interventions: Diagnostic Test: Buccal Schirmer Test

INTERVENTIONS:
Diagnostic Test: Buccal Schirmer Test — For each group, we will perform:
  * SF measurement
  * Buccal Schirmer test (BST) .

SUMMARY:
Xerostomia is a common and very bothersome manifestation that impairs the quality of life in Sjogren's syndrome. Its diagnosis mainly relies on the measurement of salivary flow (SF). Performing this test is unpleasant for the patient, lacks precision, can be influenced by certain conditions, and requires good patient cooperation. Other alternatives such as the buccal Schirmer test can be used. The aim of this study is to demonstrate the non-inferiority of the buccal Schirmer test compared to SF measurement. This is a diagnostic study comparing a group of patients (n=90) with Sjogren's syndrome (SS) and normal SF (≥0.1 ml/minute) to a group of patients with SS and decreased SF (<0.1 ml/minute).

DETAILED DESCRIPTION:
Introduction:

Xerostomia or dry mouth is a manifestation encountered in various physiological or pathological conditions. One of its main causes is Sjogren's syndrome, an autoimmune disease not specific to an organ, characterized by lymphoplasmacytic infiltration of autoimmune origin affecting mainly the salivary and lacrimal glands.

It is a debilitating condition leading to a significant impairment in quality of life primarily due to the dry mouth syndrome. Apart from the risk of corneal perforation caused by xerophthalmia, xerostomia is characterized by difficulty in chewing, swallowing especially dry foods, and speech. It is also associated with a risk of caries, dental decay, and fungal infections. Salivary flow measurement (SF) is the diagnostic method used to confirm xerostomia if it is less than 0.1 ml/minute. However, it is a test that is poorly accepted by the patient, lacks precision, can be influenced by test conditions, requires good patient cooperation, and is unpleasant for the healthcare provider.

The aim of our study is to demonstrate the non-inferiority of the buccal Schirmer test (BST) compared to SF measurement in patients with Sjogren's syndrome.

1. Objectives:

   Primary objective: Calculation of sensitivity (Se), specificity (Sp), negative predictive value (NPV), and positive predictive value (PPV) of the BST test compared to SF measurement.
2. Clinical trial design:

   2.1. Study design:

   This is a diagnostic study comparing 2 groups:
   * Group 1: consisting of 90 patients with SS and confirmed xerostomia by SF measurement (<0.1 ml/minute).
   * Group 2: consisting of 90 patients with SS and normal SF (≥0.1 ml/minute). 2.2. Inclusion and exclusion criteria: • Inclusion criteria:

   Included patients meet the following criteria:
   * age over 18 years
   * diagnosis of Sjogren's syndrome meeting the ACR/EULAR 2016 criteria. • Exclusion criteria:

   These include:
   * Cognitive or dementia disorders
   * Pregnancy 2.3. Patient allocation:

   Patients meeting the inclusion criteria will be allocated to 2 groups based on SF:
   * Group 1: patients with SF <0.1 ml/minute
   * Group 2: patients with SF ≥0.1 ml/minute. 2.4. Interventions:

   For each group, we will perform (Figure 1) :
   * SF measurement: This is the gold standard in diagnosing xerostomia. This test involves instructing the patient to collect saliva in the morning without prior stimulation (no smoking, chewing gum, or alcohol one hour before) in a graduated tube for 15 minutes. The patient should be comfortably seated with the head slightly tilted forward and mouth open to let the saliva flow. A value less than 0.1 ml/minute indicates xerostomia.
   * Buccal Schirmer test (BST) : It involves a strip of Whatman paper (blotting paper) placed in a polyethylene bag, with the first 5 mm of the strip protruding from one end of the bag. This end is then folded and placed under the patient's tongue in contact with the floor of the mouth for 5 minutes. The patient should be in a forward-leaning position, hands on knees, and eyes closed. After five minutes, the strip is removed, and the soaked part is measured in centimeters. A value <5 mm is considered pathological.

   Figure 1 : Study's flow chart
3. Data collection methods:

   Epidemiological and clinical data will be collected through interviews and data extracted from medical records.

   Epidemiological data include: age, gender, medical history such as diabetes, chronic viral infection (HCV/HIV), medications taken, previous radiotherapy, previous organ transplant, smoking, alcohol consumption.

   Clinical data include: xerophthalmia, parotid hypertrophy, cutaneous xerosis, vaginal dryness, pulmonary involvement, renal involvement, central and peripheral neurological involvement.

   All these data will be entered using the SPSS software.
4. Statistical analysis:

   It will be conducted using the SPSS software, which will allow us to obtain the contingency table as shown in Table 1.

   Table 1 : Contingency table SF

   BST + -
   * F1 F2

     * F3 F4

   This table will be used to calculate:
   * Sensitivity (Se) corresponds to the ratio: F1/(F1+F3)
   * Specificity (Sp) corresponds to the ratio: F4/(F4+F2)
   * Positive predictive value (PPV) corresponds to the ratio: F1/(F1+F2)
   * Negative predictive value (NPV) corresponds to the ratio: F4/(F4+F3)
   * Positive likelihood ratio (PLR) corresponds to the ratio: Se/(1-Sp)
   * Negative likelihood ratio (NLR) corresponds to the ratio: (1-Se) /Sp
5. Ethics and informed consent:

   Informed consent will be obtained before inclusion in the study. The patient must sign a consent form (appendix 1) after being explained in a comprehensible and simple language about the trial (appendix 2).

   This protocol will be submitted for approval to the ethics committee of the La Rabta University Hospital.

   Numbers will be assigned to patients according to their order of inclusion. This number will be used for data entry to protect patient confidentiality.
6. Funding and conflicts of interest:

The buccal Schirmer tests and the necessary equipment for FS measurement will be funded by the investigator.

All authors declare no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Included patients meet the following criteria:
* age over 18 years
* diagnosis of Sjogren's syndrome meeting the ACR/EULAR 2016 criteria.

Exclusion Criteria:

* These include:
* Cognitive or dementia disorders
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients meet the following criteria:
  * age over 18 years
  * diagnosis of Sjogren's syndrome meeting the ACR/EULAR 2016 criteria. • Exclusion criteria:
  These include:
  * Cognitive or dementia disorders
  * Pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-08-19 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 30 minutes
  ratio of the number of patients with SF+ and BST+ by the number of patients with SF+
Specificity | 30 minutes
  ratio of the number of patients with BST- and SF- by the number of patients with SF-
Positive predictive value | 30 minutes
  ratio of the number of patients with SF+ and BST+ by the number of patients with BST+
Negative predictive value | 90 minutes
  ratio of the number of patients with BST- and SF- by the number of patients with BST-

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Saïd, Principal Investigator — Centre Hospitalo-Universitaire La Rabta

IPD SHARING:
Plan to Share IPD: No
it is a diagnostic observational study. There are not many patient data collected